CLINICAL TRIAL: NCT02282852
Title: Randomised Comparison of a Standard Protocol Using Metoclopramide Versus a Hand Held Magnet to Enhance Gastric Emptying of the Small Bowel Capsule.
Brief Title: Can Steerable Capsule Endoscopy Enhance Gastric Emptying?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: STH17268
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2014-10

CONDITIONS: Patients Attending Hospital for Small Bowel Endoscopy
MeSH Terms: interventions — Capsule Endoscopy; Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wireless Capsule Endoscopy (Experimental): Wireless capsule endoscopy is the investigation modality of choice for suspected diseases of the small bowel. A small pill-sized capsule contianing a camera is swallowed by the patient. The procedure is safe and non-invasive. Normally, the pill camera travels through the gut an exits the bowel via natural means. In a small number of cases the capsule is maintained. If the capsule is still in the stomach, mobilisation is encouraged followed by an intramuscular pro-kinetic injection if this fails.
  Interventions: Device: Wireless Capsule Endoscopy
- Magnetically steerable capsule endoscopy (Active Comparator): A handheld magnet (manufactured by Intromedic Ltd.) has been developed to allow some control of the pill camera (that contains a small amount of magnetic material) in the upper GI tract. We propose that this could be used, alongside positional changes, to expedite capsule transit through the stomach thus improving completion rates and avoiding the risks of unnecessary medication.
  Interventions: Device: Magnetically steerable capsule endoscopy

INTERVENTIONS:
Device: Wireless Capsule Endoscopy
  Other Names: Swallowable pill camera
  Arms: Wireless Capsule Endoscopy
Device: Magnetically steerable capsule endoscopy
  Arms: Magnetically steerable capsule endoscopy

SUMMARY:
Small bowel wireless capsule endoscopy is the investigation modality of choice for suspected diseases of the small bowel. The procedure is safe and noninvasive, the main risk being capsule retention occurring in approximately 2% of procedures. Other problems such as incomplete examinations occur in 10-20% of procedures. Reasons include delayed gastric emptying, slow small bowel transit, faulty equipment and poor bowel preparation.

Some protocols identify the capsule position 30 minutes after ingestion using a 'realtime' viewer. If the capsule remains in the stomach, mobilisation is encouraged followed by an intramuscular prokinetic injection if this fails. This approach has disadvantages since an intramuscular injection is uncomfortable for patients. Additionally metoclopramide, commonly used for this purpose, has a risk of acute dystonic reactions particularly in young patients.

Recently a handheld magnet (Intromedic Ltd.) has been developed to enable control of the capsule in the upper GI tract. We propose that this could be used, alongside positional changes, to expedite capsule transit through the stomach thus improving completion rates and avoiding the risks of unnecessary medication. We wish to undertake a randomised controlled study comparing a standard protocol for small bowel capsule endoscopy against a hand held magnet and positional change protocol to enhance gastric emptying of the wireless capsule.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or over
* Patients attending hospital for small bowel endoscopy examination

Exclusion Criteria:

* Patients under the age of 20 years
* Patients with a permanent pacemaker, or implantable cardioverter-defibrillator
* Patients with any electronic/magnetic/mechanically controlled devices
* Patients that are pregnant
* Patients who are unable to understand or speak English

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Completion rate of small bowel endoscopy examination | Baseline
Duration of time taken for camera capsule to enter duodenum. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mark McAlindon, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom